CLINICAL TRIAL: NCT02471833
Title: Health Evaluation in African Americans Using RAS Therapy
Acronym: HEART
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Whitney Wharton, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00080192; 1RF1AG051514 (NIH)
Record Dates: First submitted 2015-06-10; First posted 2015-06-15 (Estimated); Results first posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer's Disease
Keywords: hypertension; prevention; family history; inflammation; blood brain barrier; amyloid
MeSH Terms: conditions — Alzheimer Disease; Hypertension; Inflammation | interventions — Telmisartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Telmisartan 20mg (Experimental): African American participants with untreated or treated hypertension and at high risk for Alzheimer's disease who are randomly assigned to receive telmisartan 20mg once a day orally.
  Interventions: Drug: Telmisartan 20mg
- Telmisartan 40mg (Experimental): African American participants with untreated or treated hypertension and at high risk for Alzheimer's disease who are randomly assigned to receive telmisartan 40mg once a day orally.
  Interventions: Drug: Telmisartan 40mg
- Placebo (Placebo Comparator): African American participants with untreated or treated hypertension and at high risk for Alzheimer's disease who are randomly assigned to receive a placebo to match telmisartan once a day orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan 20mg — Participants will be given 20 mg of telmisartan to be taken orally once a day before bedtime, for a duration of 8 months.
  Other Names: Micardis
  Arms: Telmisartan 20mg
Drug: Telmisartan 40mg — Participants will be given 40 mg of telmisartan to be taken orally once a day before bedtime, for a duration of 8 months.
  Other Names: Micardis
  Arms: Telmisartan 40mg
Drug: Placebo — Participants will be given placebo to be taken orally once a day before bedtime, for a duration of 8 months.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if telmisartan, an FDA approved blood pressure medication, may also have beneficial effects on Alzheimer's disease prevention in African Americans, who are at high risk for Alzheimer's disease.

DETAILED DESCRIPTION:
This study will assess if telmisartan, an FDA approved blood pressure medication, may also have beneficial effects on Alzheimer's disease (AD) prevention in African Americans, who are at high risk for Alzheimer's disease. Blood pressure medications known as angiotensin-receptor blockers have been associated with reduced risk of Alzheimer's in Caucasians because they act on the renin-angiotensin system (RAS), a key regulator of blood pressure in the body and the brain. The drugs appear to slow the progression of the disease by affecting flow of blood and the amount of plaque in the brain, but these benefits have not been tested in African Americans. The investigator will evaluate if telmisartan is able to influence the renin-angiotensin system in the brain and produce favorable effects on brain blood flow and enzymes that cause the brain plaques in Alzheimer's disease.The investigator will assess the mechanism by which telmisartan modifies the brain renin angiotensin system, cerebrospinal fluid amyloid-β, cerebral blood flow (CBF) and inflammatory markers in hypertensive African Americans.

ELIGIBILITY:
Inclusion Criteria:

* Mean resting systolic blood pressure ≥ 110 mmHg and ≤ 170 mmHg
* Family history of Alzheimer's disease
* African American

Exclusion Criteria:

* Currently in another investigational drug study
* Potassium >5.0 meq/dL at baseline
* Creatinine >1.99 mg/dL at baseline
* History of stroke or transient ischemic attack (TIA)
* Dementia
* Current use of a RAS acting medication
* Contraindication for lumbar puncture or magnetic resonance imaging
* Heart failure
* Diabetes Types I and II
* Pregnant or nursing women

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Whitney, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wharton W, Goldstein FC, Tansey MG, Brown AL, Tharwani SD, Verble DD, Cintron A, Kehoe PG. Rationale and Design of the Mechanistic Potential of Antihypertensives in Preclinical Alzheimer's (HEART) Trial. J Alzheimers Dis. 2018;61(2):815-824. doi: 10.3233/JAD-161198. PMID 29254080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Wesley Woods Health Center, Emory Alzheimer's Clinical Research Unit (ACRU), and the Emory Brain Health Center in Atlanta, Georgia, USA. Participant enrollment began April 2015 and all follow-up assessments were completed by April 15, 2022.
Groups:
- Telmisartan 20mg: African American participants with untreated or treated hypertension and at high risk for Alzheimer's disease (AD) who were randomly assigned to receive 20 mg of telmisartan to be taken orally once a day before bedtime, for a duration of 8 months.
- Telmisartan 40mg: African American participants with untreated or treated hypertension and at high risk for Alzheimer's disease who were randomly assigned to receive 40 mg of telmisartan to be taken orally once a day before bedtime, for a duration of 8 months.
- Placebo: African American participants with untreated or treated hypertension and at high risk for Alzheimer's disease who were randomly assigned to receive a placebo to match telmisartan to be taken orally once a day before bedtime, for a duration of 8 months.
Period: Overall Study
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Started | 19 | 18 | 24
Completed 8 Months of Study Treatment (Four participants in the Telmisartan 20mg group, 1 participant in the Telmisartan 40mg group, and 2 participants in the Placebo group were withdrawn from study medication prior to completing 8 months of treatment. These participants attended the Month 8 study visit and are considered as completing the study.) | 12 | 16 | 17
Completed | 16 | 17 | 19
Not Completed | 3 | 1 | 5
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Telmisartan 20mg: African American participants with untreated or treated hypertension and at high risk for Alzheimer's disease who were randomly assigned to receive 20 mg of telmisartan to be taken orally once a day before bedtime, for a duration of 8 months.
- Total: Total of all reporting groups
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo | Total
Number analyzed (Participants) | 19 | 18 | 24 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.79 (8.85) | 60.44 (7.48) | 60.54 (8.65) | 59.66 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 19. | 51
  Male | 3 | 2 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 18 | 24 | 61
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 19 | 18 | 24 | 61
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 18 | 24 | 61

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Angiotensin Converting Enzyme (ACE 1)
Description: The cerebrospinal fluid renin-angiotensin system (RAS) was assessed by measuring levels of angiotensin metabolites in a 1 milliliter (mL) sample of cerebrospinal fluid (CSF). ACE 1 helps to regulate blood pressure by converting angiotensin I to angiotensin II.
Time Frame: Baseline, Month 8
Population: This analysis includes participants who completed 8 months of study treatment, attended the Month 8 study visit, and had a sufficient sample of CSF collected. The amount of CSF collected fluctuated and some samples were not of adequate quantity to be used for every lab measurement. In some cases, participants had an unsuccessful or inadequate lumbar puncture at Baseline and then had a successful lumbar puncture at the Month 8 visit.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 10 | 15 | 16
ng/mL
  Baseline | 4043.15 (1425.34) | 4028.17 (1509.02) | 3836.31 (1627.50)
  Month 8: number analyzed (Participants) | 7 | 12 | 12
  Month 8 | 3305.21 (764.54) | 4102.96 (1498.07) | 3696.71 (1309.61)

2. Primary Outcome: Concentration of Angiotensin Converting Enzyme 2 (ACE 2)
Description: The cerebrospinal fluid renin-angiotensin system (RAS) was assessed by measuring levels of angiotensin metabolites in a 1 milliliter (mL) sample of cerebrospinal fluid (CSF). ACE 2 regulates levels of circulating angiotensin II. ACE 2 increases during illness and with Alzheimer's disease.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 14 | 16
ng/mL
  Baseline | 889.06 (870.83) | 566.43 (700.13) | 783.72 (998.95)
  Month 8: number analyzed (Participants) | 7 | 12 | 12
  Month 8 | 231.86 (47.66) | 274.17 (84.74) | 264.83 (109.40)

3. Primary Outcome: Cerebrospinal Fluid Amyloid β40
Description: Levels of amyloid β40 (Aβ40) in the cerebrospinal fluid were measured using LUMIPULSE® technology. The relationship between Aβ40 is non-linear with moderate levels showing the highest risk of future cognitive decline in some studies.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 11 | 13 | 16
picograms per milliliter (pg/mL)
  Baseline | 7704.82 (2237.94) | 9121.62 (3174.21) | 8259.13 (2176.62)
  Month 8: number analyzed (Participants) | 9 | 12 | 12
  Month 8 | 8011.44 (2688.34) | 8820.08 (2514.47) | 8300.67 (2623.31)

4. Primary Outcome: Levels of Cerebrospinal Fluid Amyloid β42
Description: Levels of amyloid β42 (Aβ42) in the cerebrospinal fluid were measured using LUMIPULSE® technology. Decreases in concentrations of amyloid β42 are indicative of a decrease in cognitive function.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 11 | 13 | 16
pg/mL
  Baseline | 611.91 (138.51) | 614.54 (193.54) | 578.31 (190.75)
  Month 8: number analyzed (Participants) | 9 | 12 | 16
  Month 8 | 620.89 (256.43) | 665.42 (278.00) | 599.25 (204.17)

5. Primary Outcome: Levels of Cerebrospinal Fluid T-tau
Description: Levels of T-tau in the cerebrospinal fluid were measured using LUMIPULSE® technology. Increases in concentrations of T-tau are indicative of a decrease in cognitive function.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 11 | 13 | 16
pg/mL
  Baseline | 347.73 (371.85) | 281.23 (89.72) | 248.94 (107.67)
  Month 8: number analyzed (Participants) | 9 | 12 | 12
  Month 8 | 393.11 (404.35) | 266.58 (83.23) | 244.58 (67.04)

6. Primary Outcome: Levels of Cerebrospinal Fluid P-tau
Description: Levels of P-tau in the cerebrospinal fluid were measured using LUMIPULSE® technology. Increases in concentrations of P-tau are indicative of a decrease in cognitive function.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 11 | 13 | 16
pg/mL
  Baseline | 29.75 (12.88) | 36.55 (11.24) | 31.58 (13.24)
  Month 8: number analyzed (Participants) | 9 | 12 | 12
  Month 8 | 30.48 (10.16) | 35.68 (13.67) | 30.48 (10.30)

7. Secondary Outcome: Interleukin-6 (IL-6) Frequency
Description: The inflammatory marker IL-6 in CSF was examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 8 | 12 | 13
pg/mL
  Baseline: number analyzed (Participants) | 7 | 12 | 13
  Baseline | 9.41 (3.25) | 10.65 (6.77) | 8.62 (3.08)
  Month 8: number analyzed (Participants) | 8 | 12 | 12
  Month 8 | 8.51 (4.73) | 8.69 (4.14) | 8.19 (3.23)

8. Secondary Outcome: Interleukin-7 (IL-7) Frequency
Description: The inflammatory marker IL-7 in CSF was examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 13 | 16
pg/mL
  Baseline | 1.88 (1.77) | 1.70 (1.57) | 1.77 (1.17)
  Month 8: number analyzed (Participants) | 8 | 12 | 12
  Month 8 | 2.06 (1.84) | 1.16 (0.66) | 1.03 (1.01)

9. Secondary Outcome: Interleukin-8 (IL-8) Frequency
Description: The inflammatory marker IL-8 in CSF was examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 13 | 16
pg/mL
  Baseline | 123.77 (64.31) | 156.99 (49.10) | 165.40 (100.25)
  Month 8: number analyzed (Participants) | 8 | 12 | 12
  Month 8 | 103.31 (42.88) | 102.11 (25.84) | 122.99 (51.36)

10. Secondary Outcome: Interleukin-9 (IL-9) Frequency
Description: The inflammatory marker IL-9 in CSF was examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 13 | 16
pg/mL
  Baseline | 96.55 (64.31) | 153.65 (71.26) | 119.18 (79.53)
  Month 8: number analyzed (Participants) | 7 | 12 | 12
  Month 8 | 81.24 (34.06) | 98.32 (28.48) | 88.22 (39.96)

11. Secondary Outcome: Interleukin-10 (IL-10) Frequency
Description: The inflammatory marker IL-10 in CSF was examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 13 | 16
pg/mL
  Baseline | 9.70 (3.31) | 11.93 (3.32) | 10.92 (3.09)
  Month 8: number analyzed (Participants) | 8 | 12 | 12
  Month 8 | 8.83 (2.31) | 10.15 (2.85) | 10.60 (2.26)

12. Secondary Outcome: Monocyte Chemoattractant Protein 1 (MCP-1) Frequency
Description: Monocyte chemoattractant protein 1 inflammatory markers in CSF were examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 13 | 16
pg/mL
  Baseline | 3369.30 (1180.22) | 3347.26 (786.79) | 3606.96 (1077.71)
  Month 8: number analyzed (Participants) | 8 | 12 | 12
  Month 8 | 2069.32 (735.75) | 2343.98 (487.36) | 2548.37 (872.88)

13. Secondary Outcome: Macrophage Derived Protein 1 (MDC-1) Frequency
Description: Macrophage derived protein 1 inflammatory markers in CSF were examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 13 | 16
pg/mL
  Baseline | 23.68 (30.61) | 13.12 (22.27) | 30.88 (67.71)
  Month 8: number analyzed (Participants) | 8 | 12 | 12
  Month 8 | 6.70 (4.84) | 9.47 (5.46) | 10.40 (4.41)

14. Secondary Outcome: Transforming Growth Factor Alpha (TGF-α) Frequency
Description: Transforming growth factor alpha inflammatory markers in CSF were examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 13 | 16
pg/mL
  Baseline | 9.42 (2.29) | 9.58 (1.65) | 9.05 (1.71)
  Month 8: number analyzed (Participants) | 8 | 12 | 12
  Month 8 | 7.56 (2.08) | 7.07 (1.61) | 7.25 (1.25)

15. Secondary Outcome: Tumor Necrosis Factor Alpha (TNF-α) Frequency
Description: Tumor necrosis factor alpha inflammatory markers in CSF were examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 13 | 16
pg/mL
  Baseline | 4.54 (4.12) | 6.72 (4.68) | 5.17 (3.28)
  Month 8: number analyzed (Participants) | 8 | 12 | 16
  Month 8 | 2.96 (0.94) | 3.12 (0.98) | 4.71 (8.63)

16. Secondary Outcome: Intercellular Adhesion Molecule 1 (ICAM-1) Frequency
Description: Intercellular adhesion molecule 1 inflammatory markers in CSF were examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 13 | 16
ng/mL
  Baseline | 207.81 (107.74) | 310.55 (258.73) | 205.18 (179.56)
  Month 8: number analyzed (Participants) | 7 | 12 | 8
  Month 8 | 472.01 (385.47) | 461.41 (290.66) | 591.69 (494.44)

17. Secondary Outcome: Vascular Cell Adhesion Molecule 1 (VCAM-1) Frequency
Description: Vascular cell adhesion molecule 1 inflammatory markers in CSF were examined.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 9 | 13 | 16
ng/mL
  Baseline | 12585.04 (10891.20) | 16838.79 (9151.95) | 13807.56 (8991.60)
  Month 8: number analyzed (Participants) | 8 | 12 | 12
  Month 8 | 12964.43 (2893.44) | 172781.50 (4513.46) | 19212.32 (8557.18)

18. Secondary Outcome: Matrix Metalloproteinase (MMP) Frequency
Description: Matrix metalloproteinase inflammatory markers will be examined in CSF.
Time Frame: Baseline, Month 8
Population: MMP was not analyzed because since developing the protocol for this study much has been learned about inflammatory cytokines and chemokines as AD preclinical biomarkers. The biological assay menu options for group analyses changed to include only those that have been shown to be related to disease state and likelihood of progression. The marker MMP was removed from the preplanned menu of inflammatory markers by the manufacturer and having MMP analyzed independently was cost prohibitive.
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Tissue Inhibitor of Metalloproteinase (TIMP) Frequency
Description: Tissue inhibitor of metalloproteinase inflammatory markers will be examined in CSF.
Time Frame: Baseline, Month 8
Population: TIMP was not analyzed because since developing the protocol for this study much has been learned about inflammatory cytokines and chemokines as AD preclinical biomarkers. The biological assay menu options for group analyses changed to include only those that have been shown to be related to disease state and likelihood of progression. The marker TIMP was removed from the preplanned menu of inflammatory markers by the manufacturer and having TIMP analyzed independently was cost prohibitive.
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: CSF-Soluble Platelet-Derived Growth Factor Receptor Beta (sPDGFRβ)
Description: Soluble Platelet-Derived Growth Factor Receptor Beta (sPDGFRβ) is a marker of breakdown in the blood brain barrier. Increased levels of sPDGFRβ indicate cognitive dysfunction.
Time Frame: Baseline, Month 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
Number analyzed (Participants) | 8 | 12 | 13
pg/mL
  Baseline: number analyzed (Participants) | 7 | 12 | 13
  Baseline | 600.30 (299.60) | 432.02 (210.85) | 403.74 (156.44)
  Month 8: number analyzed (Participants) | 8 | 12 | 12
  Month 8 | 470.93 (104.50) | 391.10 (151.23) | 471.60 (190.34)

21. Other Pre Specified Outcome: Change in Structural Magnetic Resonance Imaging and White Matter Hyperintensities
Description: High-resolution anatomical images will be acquired using a 3D-Fast Spoiled Gradient Recalled Echo (FSPGR) Sequence. White Matter Hyperintensities (WMH) will be identified by a 3D T2 Fluid Attenuated Inversion Recovery (FLAIR) Fast Spin Echo sequence. The images will be co-registered using a within-subject inter-modal alignment between structural and perfusion images. T1-weighted Spoiled Gradient Recalled (SPGR) images will be used to identify cerebrospinal fluid and white and gray matter. Increased volumes of white matter hyperintensities indicate impaired cognitive function.
Time Frame: Baseline, Month 8
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Change in Arterial Spin Labeling-Magnetic Resonance Imaging
Description: Echoplanar T1 mapping scans will be used for image registration and a scout image of the head will be obtained in order to choose the appropriate location for spin labeling and flow imaging. Arterial Spin Labeling images will be acquired using a custom 3D stack of interleaved spirals fast spin echo sequences and will be averaged in order to improve the signal-to-noise ratio. Images will be interpolated and smoothed in a panel by using a 0.5-pixel, full-width, half-maximum Gaussian kernel. Regional perfusion will be quantified in each hemisphere and maps of cerebral vasoreactivity will be obtained by co-registration of perfusion and anatomical images.
Time Frame: Baseline, Month 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the baseline assessment and continued through the final assessment at Month 8.
Description: Participants were asked if they had experienced specific, anticipated adverse events. There was also a field for reporting other adverse events that were not specified.
Arm/Group | Telmisartan 20mg | Telmisartan 40mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18 | 0/24
Other Adverse Events (participants affected / at risk) | 13/19 | 13/18 | 15/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 20mg (N=19) | Telmisartan 40mg (N=18) | Placebo (N=24)
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 2
Excessive swelling (General disorders) | 1 | 0 | 2
Hypotension (Cardiac disorders) | 2 | 0 | 0
Postural hypotension (Cardiac disorders) | 1 | 2 | 1
Persistent cough (General disorders) | 4 | 1 | 1
Dizziness (General disorders) | 3 | 2 | 2
Angina pectoris (Cardiac disorders) | 1 | 0 | 2
Angioedema (Cardiac disorders) | 1 | 0 | 0
Nausea/vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Syncope (General disorders) | 0 | 0 | 0
Vertigo (General disorders) | 3 | 1 | 0
Abnormal kidney function (Renal and urinary disorders) | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 8 | 2 | 1
Unusual muscle aches (Musculoskeletal and connective tissue disorders) | 7 | 5 | 3
Fatigue (General disorders) | 2 | 1 | 0
Sore throat (General disorders) | 1 | 0 | 0
Headache (General disorders) | 1 | 1 | 2
Dry mouth (General disorders) | 1 | 2 | 0
Night sweats (General disorders) | 1 | 0 | 0
Out of range labs (General disorders) | 1 | 0 | 0
Cold symptoms (Infections and infestations) | 0 | 1 | 0
Increased body temperature (General disorders) | 0 | 0 | 1
Acid reflux (Gastrointestinal disorders) | 0 | 0 | 1
Trouble falling asleep (General disorders) | 0 | 0 | 1
Indigestion (Gastrointestinal disorders) | 0 | 0 | 1
Difficulty swallowing (General disorders) | 0 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Heart palpitations (Cardiac disorders) | 0 | 0 | 1
Low energy (General disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Weight loss (General disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Unanticipated expenses related to the Coronavirus Disease 2019 (COVID-19) pandemic resulted in less funds toward the end of this study impacting the post processing of neuroimaging scans.The researchers are submitting for additional funding for imaging processing and analyses, as well as searching for an expert who is available to perform imaging processing. Results for the magnetic resonance imaging outcomes will be reported as soon as possible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT02471833/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/33/NCT02471833/ICF_000.pdf